CLINICAL TRIAL: NCT02324608
Title: A Pilot Study of Neoadjuvant Cetuximab in Advanced Squamous Cell Carcinomas of Skin (SCCS)
Brief Title: Cetuximab Before Surgery in Treating Patients With Aggressive Locally Advanced Skin Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Rutgers Cancer Institute of New Jersey (Other)
Responsible Party: Principal Investigator, Adam Berger, MD, Principal Investigator, Rutgers Cancer Institute of New Jersey
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 091303; NCI-2014-02027 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); Pro20140000555 (Other: Rutgers Cancer Institute of New Jersey); P30CA072720 (NIH)
Record Dates: First submitted 2014-10-28; First posted 2014-12-24 (Estimated); Results first posted 2023-12-20 (Actual); Last update posted 2023-12-20 (Actual); Status verified 2023-11

CONDITIONS: Recurrent Skin Cancer; Squamous Cell Carcinoma of the Skin
MeSH Terms: conditions — Skin Neoplasms | interventions — Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (cetuximab) (Experimental): Patients receive cetuximab IV over 60-120 minutes once weekly for 8 weeks.
  Interventions: Biological: cetuximab; Other: laboratory biomarker analysis

INTERVENTIONS:
Biological: cetuximab — Given IV
  Other Names: C225; C225 monoclonal antibody; IMC-C225; MOAB C225; monoclonal antibody C225
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This pilot clinical trial studies the side effects and how well cetuximab before surgery works in treating patients with skin cancer that forms, grows, and spreads quickly and has spread from where it started to nearby tissue or lymph nodes. Monoclonal antibodies, such as cetuximab, may block tumor growth in different ways be targeting certain cells. Giving cetuximab before surgery may make the tumor smaller and reduce the amount of normal tissue that needs to be removed.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the response rate of cetuximab by Response Evaluation Criteria in Solid Tumors (RECIST) criteria in patients with advanced squamous cell carcinoma of skin (SCCS).

II. To assess whether neoadjuvant cetuximab given in this patient population is both safe and feasible.

SECONDARY OBJECTIVES:

I. To measure the progression free and overall survival of patients with advanced SCCS who receive neoadjuvant cetuximab.

II. To determine the conversion to resectability of patients treated with neoadjuvant cetuximab and capture changes in reconstructive options rendered possible by neoadjuvant treatment.

III. Analyze the relationship of known deoxyribonucleic acid (DNA) mutations in tumor per the FoundationOneTM genomic profile, and correlate to clinical endpoints such as clinical benefit and conversion to resectability to discover potential markers of response and/or resistance.

IV. Measure the downstream activation of signaling pathways without a known driver, including the epidermal growth factor receptor (EGFR) pathway.

V. Determine if tumor shrinkage with cetuximab is associated with increased apoptosis as evidenced by activated caspase-3, in pre- and post- treatment tumor tissues.

VI. Determine whether cetuximab results in increased antibody-dependent cell cytotoxicity (ADCC) in post-, compared with pre-treatment tumor tissues.

OUTLINE:

Patients receive cetuximab intravenously (IV) over 60-120 minutes once weekly for 8 weeks.

After completion of study treatment, patients are followed up every 3 months for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have untreated or relapsed SCCS that is considered to be aggressive and locally advanced by the following criteria: tumors 2 cm or more, tumors invading deep tissues such as muscle, cartilage or bone; tumors showing perineural invasion, and/or tumors metastatic to loco-regional lymph nodes; patients may have had prior surgical interventions or been treated with investigational agents with residual or recurrent disease
* Patients must give informed consent
* Patients must agree to pre- and post-treatment biopsies
* Patients must have an Eastern Cooperative Oncology Group (ECOG) performance status =< 2
* Estimated life expectancy of at least 12 weeks
* Negative pregnancy test

Exclusion Criteria:

* Second primary malignancy only if treatment would interfere with the patient's participation in this trial in the opinion of the treating physician; clear exceptions are 1) patient had a second primary malignancy but has been treated and disease free for at least 3 years, 2) in situ carcinoma (e.g. in situ carcinoma of the cervix) and, 3) additional skin cancers that have been definitively treated by surgery and/or radiation; patients with chronic lymphocytic leukemia will be allowed if their blood counts are within acceptable hematologic parameters and if they are not currently requiring cytotoxic or biologic anticancer treatment (supportive treatment such as intravenous immunoglobulin [IVIG] is permitted)
* Patients with distant organ metastases will not be included in this study
* Serious concomitant systemic disorders (including active infections) that would compromise the safety of the patient or compromise the patient's ability to complete the study, at the discretion of the investigator
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to cetuximab or other agents used in the study
* Women who are pregnant; women of childbearing age must agree to undergo a pregnancy test prior to therapy and to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation and for 6 months after; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately
* Serum calcium (ionized or adjusted for albumin) < 8 mg/dl (1.75 mmol/L) or > 12.5 mg/dl (> 3.1 mmol/L) despite intervention to normalize levels
* Magnesium < 1.4 mg/dl (< 0.4 mmol/L) or > 3 mg/dl (> 1.23 mmol/L) despite intervention to normalize levels
* Potassium < 3.5 mmol/L or > 6 mmol/L despite intervention to normalize levels
* Prior radiation therapy is not an exclusion however, patient must have documented progression at the radiation site

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2015-01-30 (Actual); Primary Completion 2020-12-09 (Actual); Study Completion 2023-05-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adam Berger, MD, Principal Investigator — Rutgers Cancer Institute of New Jersey
Locations (1):
- Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Cetuximab)
Started | 15
Completed | 15
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Cetuximab)
Number analyzed (Participants) | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 12
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 15
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 15
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Response Rate of Cetuximab by RECIST Criteria
Description: A one-sided Binomial exact test will be used.
Time Frame: Up to 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Cetuximab)
Number analyzed (Participants) | 15
Participants | 15

2. Secondary Outcome: Progression-free Survival
Description: The estimation of progression-free survival will be performed by the Kaplan-Meier product limit method. Descriptive statistics for all outcome measures will be provided. To evaluate the association between variables, either chi-square test (categorical vs. categorical) or two sample t-test (categorical vs. continuous) or correlation (continuous vs. continuous) will be used depending upon the types of variables in comparison.
Time Frame: Up to 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Cetuximab)
Number analyzed (Participants) | 15
Participants | 4

3. Secondary Outcome: Overall Survival
Description: The estimation of overall survival will be performed by the Kaplan-Meier product limit method. Descriptive statistics for all outcome measures will be provided. To evaluate the association between variables, either chi-square test (categorical vs. categorical) or two sample t-test (categorical vs. continuous) or correlation (continuous vs. continuous) will be used depending upon the types of variables in comparison.
Time Frame: Up to 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Cetuximab)
Number analyzed (Participants) | 15
Participants | 8

4. Secondary Outcome: Downstream Activation of Signaling Pathways Without a Known Driver, Including the EGFRpathway
Description: Measure the downstream activation of signaling pathways without a known driver, including the EGFRpathway
Time Frame: Up to 2 years
Population: no data collected
Arm/Group | Treatment (Cetuximab)
Number analyzed (Participants) | 0

5. Secondary Outcome: Potential Markers of Response and/or Resistance to Cetuximab Therapy
Description: Analyze the relationship of known DNA mutations in tumor per the FoundationOneTM genomic profile, and correlate to clinical endpoints such as clinical benefit and conversion to resectability to discover potential markers of response and/or resistance to cetuximab therapy.
Time Frame: Up to 2 years
Population: no data collected
Arm/Group | Treatment (Cetuximab)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Up to 2 years after the last participant receives treatment.
Arm/Group | Treatment (Cetuximab)
All-Cause Mortality (participants affected / at risk) | 8/15
Serious Adverse Events (participants affected / at risk) | 2/15
Other Adverse Events (participants affected / at risk) | 15/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Cetuximab) (N=15)
Ear pain (Ear and labyrinth disorders) | 1 (1)
Lung infection (Infections and infestations) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Cetuximab) (N=15)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 6 (7)
Rash acneiform (Skin and subcutaneous tissue disorders) | 5 (8)
Dry skin (Skin and subcutaneous tissue disorders) | 3 (3)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1 (1)
Hypomagnesemia (Metabolism and nutrition disorders) | 9 (10)
Dehydration (Metabolism and nutrition disorders) | 2 (2)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Chills (Gastrointestinal disorders) | 1 (1)
Pain (General disorders) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 2 (2)
Bruising (Injury, poisoning and procedural complications) | 1 (1)
Wound complication (Injury, poisoning and procedural complications) | 1 (1)
Hypertension (Vascular disorders) | 3 (6)
Hypotension (Vascular disorders) | 1 (1)
Eye disorders - Other, specify (Eye disorders) | 2 (2)
Dry eye (Eye disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 2 (2)
Abdominal distension (Gastrointestinal disorders) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 1 (1)
Esophageal pain (Gastrointestinal disorders) | 1 (1)
Oral pain (Gastrointestinal disorders) | 1 (1)
Rash pustular (Infections and infestations) | 2 (9)
Lung infection (Infections and infestations) | 1 (1)
Alkaline phosphatase increased (Investigations) | 1 (1)
Creatinine increased (Investigations) | 1 (1)
Weight loss (Investigations) | 1 (1)
Headache (Nervous system disorders) | 2 (2)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (2)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 1 (1)
Ear and labyrinth disorders - Other, specify (Ear and labyrinth disorders) | 1 (3)
Ear pain (Ear and labyrinth disorders) | 1 (1)
Vaginal discharge (Reproductive system and breast disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-01-24): https://cdn.clinicaltrials.gov/large-docs/08/NCT02324608/Prot_SAP_000.pdf
  • Informed Consent Form (2020-01-24): https://cdn.clinicaltrials.gov/large-docs/08/NCT02324608/ICF_001.pdf